CLINICAL TRIAL: NCT06292351
Title: Multicenter Randomized Double-blind Placebo-controlled Three-arm Parallel-group Clinical Study to Evaluate the Efficacy and Safety of DMB-I in the Treatment of Dementia Associated With Alzheimer's Disease
Brief Title: DMB-I in the Treatment of Alzheimer Type Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bigespas LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMBN_ALZH-2022-II
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease; Dementia of Alzheimer Type
MeSH Terms: conditions — Alzheimer Disease | interventions — latrepirdine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- DMB-I (Dimebon) + Placebo (Experimental)
  Interventions: Drug: DMB-I (Dimebon); Other: Placebo
- DMB-I (Dimebon) (Experimental)
  Interventions: Drug: DMB-I (Dimebon)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DMB-I (Dimebon) — 20 mg 3 times a day, or 10 mg + 10 mg 3 times a day (for DMB-I + Placebo arm)
  Arms: DMB-I (Dimebon); DMB-I (Dimebon) + Placebo
Other: Placebo — 20 mg 3 times a day, or 10 mg + 10 mg 3 times a day (for DMB-I + Placebo arm)
  Arms: DMB-I (Dimebon) + Placebo; Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of DMB-I for the treatment of patients with Alzheimer type dementia.

DETAILED DESCRIPTION:
This is a multicenter, randomized, placebo-controlled study that is to assess efficacy and safety, to select the optimal therapeutic dose of the drug and to test the hypothesis of superiority of DMB-I (Dimebon) over placebo in patients with mild to moderate Alzheimer's disease.

The study is planned to be conducted in clinical sites of the Russian Federation.

Patients meeting all the eligibility criteria will be randomized into one of three treatment arms:

1. DMB-I (Dimebon) 1 tab + Placebo 1 tab 3 times a day.
2. DMB-I (Dimebon) 2 tab 3 times a day.
3. Placebo 2 tab 3 times a day.

The total study duration for each patient is approximately 182 days broken down as follows:

Screening period: up to 14 days, Treatment period: 26 weeks, Follow-up period: 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent to participate in the study.
2. Patients of any gender aged 60 to 90 years inclusive.
3. Patients diagnosed with mild to moderate Alzheimer type dementia according to the NINCDS-ADRDA criteria, receiving basic treatment with memantine at a daily dose of 20 mg for at least 2 months.
4. The MMSE score is in the range of 10-23 inclusive.
5. No signs of dementia of vascular origin according to CT/MRI data. Repeated Acute Cerebrovascular Accidents (focal infarctions) in brain areas that are critical for cognitive functions and behavior are the mandatory neuroimaging signs of vascular dementia.
6. The presence of a caregiver who is in contact with the patient a significant part of the time, agrees to accompany the patient to all visits, monitor the intake of the study drug and fill out the patient's diary.
7. Patients who are able to undergo the tests provided for in the protocol.

Exclusion Criteria:

1. Patients diagnosed with other diseases that cause dementia (severe hypothyroidism, anemia, brain tumor, including a history of neuroinfections, etc.) according to medical history, medical documentation and the results of additional examination methods.
2. History of other neurodegenerative diseases of the brain, Parkinson's disease, multiple sclerosis, demyelinating diseases of the nervous system, hereditary degenerative diseases of the central nervous system, abnormalities of the nervous system, uncontrolled epilepsy, hallucinations, other neurological disorders seriously affecting motor or cognitive function, in the opinion of the investigator.
3. History of intolerance to any of the components of the study drug.
4. History of stroke.
5. Active oncological process.
6. The need for surgeries on the vessels of the neck or brain, including endovascular interventions, during the study.
7. Signs of significant uncontrolled concomitant disease that, in the opinion of the Investigator, could prevent the patient from participating in the study, including:

   * Respiratory system disorders;
   * Cardiovascular system disorders;
   * Severe renal impairment (glomerular filtration rate <30ml/min);
   * Severe liver dysfunction (ALT, AST > 2 times the upper limit of normal);
   * Endocrine system disorders;
   * Gastrointestinal disorders.
8. Systemic autoimmune diseases or vascular collagenoses requiring previous or current treatment with systemic drugs.
9. Use of drugs that negatively affect cognitive function (tricyclic antidepressants, benzodiazepines, antipsychotics, hypnotics, etc.), as well as drugs of prohibited therapy (including Cerebrolysin, preparations of ginkgo biloba extract, any other drugs with nootropic, antioxidant, metabolic effects, as well as drugs used to treat dementia). Situational use of psychotropic drugs (e.g., for the treatment of insomnia, or to relieve agitation and anxiety) is permitted
10. Moderate to severe depression (Hamilton scale score of 14 or more).
11. Smoking.
12. Episodes of alcohol or drug abuse within the last 6 months.
13. Inability to comply with study procedures even with the assistance, in the opinion of the investigator.
14. Episodes of other serious or unstable neurological, metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal or urological disorders.
15. Myocardial infarction within 12 months prior to screening.
16. Known systemic infection (viral hepatitis, HIV, tuberculosis, syphilis).
17. Life expectancy less than 26 weeks after randomization.
18. Men of reproductive potential who are unwilling to use adequate contraceptive methods.
19. Participation in another clinical trial within the last 6 months.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2023-12-27 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Mean change in Alzheimer's Disease Assessment Scale score after 26 weeks of therapy (Visit 6) compared to baseline (Visit 0) in patients receiving the study drug or placebo | Baseline (Visit 0) and 26 weeks (Visit 6)
  The scale's minimum score - 0, maximum score - 82, where the higher score means the worse outcome

SECONDARY OUTCOMES:
Mean change in cognitive impairment score on the Alzheimer's Disease Assessment Scale after 12 weeks of therapy compared to baseline | Baseline (Visit 1) and 12 weeks of therapy (Visit 4)
  The scale's minimum score - 0, maximum score - 82, where the higher score means the worse outcome
Mean change in Mini-Mental State Examination score after 12 weeks of therapy (Visit 4) and after 26 weeks of therapy (Visit 6) compared to baseline (Visit 0) | Baseline (Visit 0), 12 weeks of therapy (Visit 4) and 26 weeks of therapy (Visit 6)
  The min/max score values are 0/30 respectively, where the higher score means the better outcome
Change in the quality of life of patients according to the Quality of Life - Alzheimer's Disease questionnaire after 12 weeks of therapy (Visit 4) and after 26 weeks of therapy (Visit 6) compared to baseline (Visit 1) | Baseline (Visit 1), 12 weeks of therapy (Visit 4) and 26 weeks of therapy (Visit 6)
  The scale has 13 items, that may be evaluated on 13-52 points, where the higher score means the better outcome
Change in the general clinical impression in accordance with the Clinical Global Impressions Scale after 12 weeks of therapy (Visit 4) and after 26 weeks of therapy (Visit 6) compared to baseline (Visit 1) | Baseline (Visit 1), 12 weeks of therapy (Visit 4) and 26 weeks of therapy (Visit 6)
  The scale consists of 3 blocks, which may be evaluated on 0 to 7 points for each of the first two blocks, and on 1 to 16 points for the third block. The higher score means the worse outcome.
Dynamics on the Lawton's Instrumental activities of daily living scale after 12 weeks of therapy (Visit 4) and after 26 weeks of therapy (Visit 6) compared to baseline (Visit 1) | Baseline (Visit 1), 12 weeks of therapy (Visit 4) and 26 weeks of therapy (Visit 6)
  The min/max score values are 0/8 respectively, where the higher score means the worse outcome

CONTACTS AND LOCATIONS:
Locations (7):
- Russia (7):
  - State autonomous healthcare institution "Transregional Clinical Diagnostic Center", Kazan'
  - Federal State Budgetary Institution "Federal center for brain and neurotechnologies" of the Federal Medical and Biological Agency (FSBI "FCBN" of Russia's FMBA), Moscow
  - Federal State Autonomous Educational Institution of Higher Education I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University), Moscow
  - State public healthcare institution Leningrad regional psychoneurologic dispensary, Roshchino
  - "Medical Center Nova Vita", Rostov-on-Don
  - Saint Petersburg State budgetary healthcare institution "City Hospital № 40 of Kurortniy district", Saint Petersburg
  - "Centre of evidence-based medicine" LLC, Yaroslavl

REFERENCES:
- See also: Differences in bioavailability and cognitive-enhancing activity exerted by different crystal polymorphs of latrepirdine (Dimebon®) — https://www.frontiersin.org/journals/pharmacology/articles/10.3389/fphar.2023.1091858/full